CLINICAL TRIAL: NCT06553781
Title: A Single-arm, Multicenter Clinical Study of Fruquintinib Combined With Cadonilimab Injection and Temozolomide in Second-line and Subsequent Treatment of Advanced Melanoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief physician of Medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2407299-2
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Temozolomide、Fruquintinib、Cadonilimab — Combination treatment period:
  Fruquintinib: 4mg d1-21, po qd q4w; Cadonilimab 6mg/kg, ivgtt q2w; Temozolomide: 150~200mg/m2, poqd, d1-5, q4W; The combined treatment lasted 6 cycles.
  Maintenance treatment:
  Fruquintinib: 4mg d1-21, po qd q4w; Cadonilimab 6mg/kg, ivgtt q2w; The maximum duration of maintenance treatment is not more than 2 years.

SUMMARY:
This single-arm, multicenter clinical study enrolled patients with advanced malignant melanoma who had failed previous first-line therapy (cutaneous melanoma patients were excluded), and patients with BRAF V600 mutations required targeted therapy.

DETAILED DESCRIPTION:
Combination treatment period:

Fruquintinib: 4mg d1-21, po qd q4w;

Cadonilimab 6mg/kg, ivgtt q2w;

Temozolomide: 150~200mg/m2, poqd, d1-5, q4W;

The combined treatment lasted 6 cycles.

Maintenance treatment:

Fruquintinib: 4mg d1-21, po qd q4w;

Cadonilimab 6mg/kg, ivgtt q2w;

The maximum duration of maintenance treatment is not more than 2 years.

The study was divided into three stages: screening period, treatment period and follow-up period. The treatment period is a treatment cycle every 4 weeks. During the treatment period, imaging methods will be used to evaluate the tumor status every 8 weeks (±7 days) until the patient's disease progresses (RECIST 1.1) or death (during the treatment of the patient) or toxicity becomes intolerable. The tumor treatment status and survival status of the patient after disease progression should be recorded.

Safety indicators include adverse events, laboratory tests, vital signs, and changes in electrocardiogram and cardiac ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Age 18-75 years old (including 18 and 75 years old), gender is not limited;
3. Stage IV melanoma determined by pathology or cytology;
4. Patients with advanced malignant melanoma who have failed previous first-line therapy (cutaneous melanoma patients are excluded) and patients with BRAF V600 mutations need to be admitted after targeted therapy.
5. 4 weeks or more since the last systematic treatment before enrollment;
6. ECOG physical condition 0-1 score;
7. Expected survival ≥3 months;
8. Must have at least one measurable lesion (RECIST version 1.1);
9. The functions of vital organs meet the following requirements (the use of any blood components and cell growth factors within 14 days prior to enrollment is not allowed) :

   Absolute neutrophil count ≥1.5×109/L;

   Platelet ≥100×109/L;

   Hemoglobin ≥90g/L;

   Total bilirubin < 1.5 ULN;

   ALT and/or AST < 1.5 times ULN;

   Serum creatinine < 1.5 ULN;

   endogenous creatinine clearance ≥50ml/min;
10. Women of childbearing age need to take effective contraceptive measures;
11. Good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Failure to comply with the study protocol or study procedure;
2. Patients with active brain metastases;
3. Received organ surgery 6 weeks before enrollment;
4. Had other malignant tumors within 5 years prior to admission, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
5. Severe cardiovascular disease, including unstable angina pectoris or myocardial infarction, in the 6 months prior to enrollment;
6. Subjects who are allergic to the investigational drug or any of its adjuncts;
7. Participated in other domestic unapproved or unmarketed drug clinical trials and accepted the corresponding experimental drug treatment within 4 weeks before enrollment;
8. International Standardized Ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN;
9. The investigator identified clinically significant electrolyte abnormalities;
10. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
11. Poorly controlled diabetes mellitus was present before enrollment (fasting glucose concentration ≥CTCAE level 2 after formal treatment);
12. Had any disease or condition affecting drug absorption before enrollment, or the patient could not take the drug orally;
13. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unresectable tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
14. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding within 3 months > 30 mL, hematemesis, stool, stool blood), hemoptysis (within 4 weeks >; 5 mL of fresh blood) or had a thromboembolic event (including stroke events and/or transient ischemic attacks) within 12 months;
15. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; New York Heart Association (NYHA) Grades for Congestive Heart Failure >Level 2; Ventricular arrhythmias requiring medical treatment; LVEF (Left ventricular Ejection Fraction) < 50%;
16. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);
17. Known human immunodeficiency virus (HIV) infection. A known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000 IU/ml) must be ruled out for a known hepatitis B virus (HBV) carrier; Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL);
18. Unmitigated toxicity higher than CTCAE v5.0 grade 1 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;
19. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
20. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 14 days before enrollment;
21. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
22. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume >1.0g;
23. The patients considered by the investigators to be unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR（objective response rate） | 5 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
OS Overall survival | two years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
DCR Disease control rate | two years
  From date of randomization until the end of treatment or the date of first documented progression or date of death from any cause, whichever came first,
PFS Progression-free survival | 5 months
  PFS were defined as from date of randomization until the date of first documented progression or date of death from any cause, whichever came first
Safety | two years
  Adverse events as assessed by NCI CTCAE v5.0overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use

IPD SHARING:
Plan to Share IPD: No